CLINICAL TRIAL: NCT05382741
Title: Study of Adjuvant Durvalumab (MEDI4736) Plus Regorafenib vs Untreated Control in Stage IV Colorectal Cancer Patients With no Evidence of Disease (NED): VIVA Trial
Brief Title: Adjuvant Durvalumab Plus Regorafenib vs Untreated Control in Stage IV Colorectal Cancer Patients With no Evidence of Disease (NED): VIVA Trial
Acronym: VIVA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ospedale Policlinico San Martino (Other)
Collaborators: Associazione Italiana per la Ricerca sul Cancro (Other); Gruppo Italiano per lo studio dei Carcinomi dell'Apparato Digerente (Other); Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VIVA TRIAL
Record Dates: First submitted 2022-05-10; First posted 2022-05-19 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Colorectal Cancer Stage IV; No Evidence of Disease State
Keywords: NED state; adjuvant; tyrosine kinase inhibitors; immunotherapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — durvalumab; regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DURVALUMAB + REGORAFENIB (Experimental): Durvalumab 1500 mg (120-minute IV infusion) every 28 days, Regorafenib 90 mg/die orally once daily for 21 days in a 28-day cycle.
  Treatment will be administred up to 1 year.
  Interventions: Drug: Durvalumab Injection for intravenous use 500 mg vial solution for infusion; Drug: Regorafenib 30 mg capsules
- CONTROL ARM (No Intervention): Observation (follow-up).
  Crossover to the experimental arm is allowed in case of relapse.

INTERVENTIONS:
Drug: Durvalumab Injection for intravenous use 500 mg vial solution for infusion — MEDI4736
  Other Names: Imfinzi
  Arms: DURVALUMAB + REGORAFENIB
Drug: Regorafenib 30 mg capsules — BAY73-4506
  Other Names: Stivarga
  Arms: DURVALUMAB + REGORAFENIB

SUMMARY:
The purpose of this study is to evaluate the efficacy of Durvalumab plus Regorafenib versus observation for patients with stage IV colorectal cancer achieving the no evidence of disease state.

The NED state can be achieved in any line of treatment and it is defined as:

1. R0 resection for surgery,
2. the complete ablation defect covering the lesion on CT scan for radiofrequency,
3. the erogation of ≥ 60 Gy for stereotactic radiotherapy,
4. complete response to antineoplastic treatments on CT scan. In all these cases CEA and CA 19.9 must be within normal limits at the time of randomization.

Participants in this study will receive:

Experimental arm:

Regorafenib 90 mg d1-21 every 28 days plus Durvalumab 1500 mg every 28 days for 1 year

Control arm:

Observation (crossover to Experimental arm is allowed in case of relapse)

Tumor assessment will be performed every 12 weeks.

DETAILED DESCRIPTION:
The safety run-in phase is planned for the first 4 patients randomized to the experimental arm using a starting dose of 60 mg/die of Regorafenib (and fixed 1500 mg of Durvalumab), to be escalated after 2 months to 90 mg/die if < 2 patients report serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years; ECOG PS 0-1;
2. Body weight >30 kg;
3. Histologically confirmed diagnosis of colorectal adenocarcinoma;
4. Patients must be in NED after completion of any treatments for stage IV CRC, including resections, RFA; RT with or without neoadjuvant/adjuvant therapies or CR after chemotherapy;
5. Patients must be randomized within 10 weeks since the achievement of the NED state. Those who have also received adjuvant therapy following the locoregional treatment are still eligible, provided they are randomized within 4 weeks since the last chemotherapy cycle;
6. NED state ascertained by means of CT scan and/or PET scan and/or MRI scan;
7. Life expectancy of at least 12 weeks;
8. CEA within normal limits;
9. No residual toxicity from previous chemotherapy;
10. Adequate organ function;

Exclusion criteria:

1. MSI/dMMR patients;
2. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia and vitiligo;
3. Active or prior documented autoimmune or inflammatory disorders;
4. Relevant concomitant comorbidities;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 182 (Estimated)
Dates: Start 2022-03-02 (Actual); Primary Completion 2024-03-02 (Estimated); Study Completion 2024-03-02 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival | approximately 48 months
  Disease free survival, defined as the time from the date of randomization to the earliest documented disease relapse (local or distant), death due to any cause or two consecutive increases of CEA above upper limit (time gap no longer than 30 days).

SECONDARY OUTCOMES:
18 months - Disease Free Survival | approximately 48 months
  Disease free survival, defined as the time from the date of randomization to the earliest documented disease relapse (local or distant), death due to any cause or two consecutive increases of CEA above upper limit (time gap no longer than 30 days).
Overall Survival | approximately 48 months
  Overall survival, defined as the time from the date of randomization to death due to any cause
Incidence of adverse events | approximately 48 months
  An adverse event was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
  Toxicity/adverse events are classified according to NCI CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Sobrero, MD, Principal Investigator — OSPEDALE SAN MARTINO IRCCS
Locations (1):
- IRCCS Ospedale Policlinico San Martino, Genoa, Liguria, Italy

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-16): https://cdn.clinicaltrials.gov/large-docs/41/NCT05382741/Prot_SAP_000.pdf